CLINICAL TRIAL: NCT07158177
Title: Clareon PanOptix Versus AcrySof PanOptix : Prospective Study Comparing Contrast Sensitivity. Study of Two Different Material of Intra Ocular Multifocal Lenses Aiming to Compare the Effect on Contrast Sensitivity.
Brief Title: Clareon PanOptix Versus AcrySof PanOptix : Prospective Study Comparing Contrast Sensitivity
Acronym: CLAYRE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Alcon Research (Industry); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: APHP241077; IDRCB (Other: 2025-A00658-41)
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Cataract and IOL Surgery
Keywords: Multifocal Intra Ocular Lens; Presbyopia Correcting Intra Ocular Lens (PCIOL).; Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clareon™ PanOptix™, toric or no-toc (Experimental)
  Interventions: Device: Clareon Panoptix
- AcrySof™ IQ PanOptix™, toric or no-toric (Active Comparator)
  Interventions: Device: Acrysof™ PanOptix™ toric or not, trifocal IOL CE marked, Alcon company.

INTERVENTIONS:
Device: Acrysof™ PanOptix™ toric or not, trifocal IOL CE marked, Alcon company. — both of the patient's eyes will be implanted: 1 CPO and the other APO
  Arms: AcrySof™ IQ PanOptix™, toric or no-toric
Device: Clareon Panoptix — both of the patient's eyes will be implanted: 1 CPO and the other APO
  Arms: Clareon™ PanOptix™, toric or no-toc

SUMMARY:
Retrospective, comparative, interventional, randomized, single-center study, contralateral (the patient's 2 eyes will be implanted: 1 CPO and the other APO) Patients presenting for cataract surgery with a request for presbyopia correction and managed as part of routine clinical practice.

The main aim of the study is to demonstrate that contrast sensitivity is better with the Clareon PanOptix (CPO) intraocular lens (IOL) compared with the AcrySof PanOptix (APO) IOL 3 months after implantation.

DETAILED DESCRIPTION:
Visit at Day3-10: usual follow-up visit, no additional examinations as part of the clinical investigation.

Visit at 1 month: usual follow-up visit, no additional examinations as part of the clinical investigation.

3-month visit (end of clinical investigation): usual follow-up visit, plus contrast vision test and non-invasive aberrometry test (I-Trace) as part of the clinical investigation.

Regarding a cataract surgery with a request for presbyopia, the protocol evaluate two differents devices (IOL intraocular lens).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age
* Patients presenting for cataract surgery in routine clinical practice and eligible for multifocal IOL implantation (toric and non-toric)
* Patients with grade 2/3 cataract density and comparable visual acuity in both eyes
* Patient with a pregnancy test (negative pregnancy test), if applicable
* Patient with signed consent to participate in the study
* Patient affiliated to a social security scheme or entitled beneficiary

Exclusion Criteria:

* Children < 18 years of age
* Pregnancy or breast-feeding in progress or planned during the study.
* History of anterior (cornea, anterior chamber, sulcus) or posterior (uveal, vitreoretinal) segment pathology, including retinal vascular occlusive disease, retinal detachment or peripheral retinal laser photocoagulation, AMD, glaucoma.
* Any inflammation of the anterior or posterior segment, whatever the etiology, and/or history of any disease with intraocular inflammatory repercussions.
* Clinically significant corneal pathology (epithelial, stromal and/or endothelial) that could have an impact on visual results.
* Clinically significant moderate or severe dry eye that could affect study measurements.
* History of intraocular or corneal surgery (refractive or trauma-related).
* Presence or history of amblyopia or monofixation syndrome.
* Subjects with conditions that increase the risk of zonular disruption during the phacoemulsification procedure that may affect the centration or postoperative orientation of the IOL.
* Any other planned eye surgery, including, but not limited to, limbal relaxing incision (LRI)/astigmatic keratotomy and laser refractive surgery (LASIK).
* Irregular astigmatism identified by corneal topography
* Patients under guardianship, curatorship or safeguard of justice, as well as pregnant or breast-feeding women (article L1121-5 of the CSP).1.1
* Patient under AME

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Contrast sensitivity measured at 3 months | 3 months
  AULCSF (Area under the log contrast sensitivity function) at different spatial frequencies (1,5 ; 3 ; 6 ; 12 cycles par degré (cpd)) in monocular vision and under mesopic condition without glare.

SECONDARY OUTCOMES:
Contrast sensitivity measured at 3 months | 3 months
  AULCSF monocular in photopic condition with and without glareat 3 months.
Uncorrected and corrected Visual acuity (UCVA and CVA) or in monocular and binocular vision at different distances (4 meters for Distance- 66 centimeters of intermediate- 40 cm for Near) | 3 months
  UDVA, UIVA, UNVA, BCDVA, DCIVA, DCNVA
Refractive stability | 1 and 3 months
  Comparison of refractive error between 1 and 3 months
OSI : Objective Scatter Index: monocular | 3 months
  Comparison of refractive error between 1 and 3 months
Glistenings | 3 months
  Using Miyata scale

CONTACTS AND LOCATIONS:
Overall Officials: Dominique MONNET, MD, PhD, Principal Investigator — Université Paris Cité, Faculté de Santé / UFR de médecine
Locations (1):
- Assistance Publique - Hôpitaux de Paris, Ophtalomopôle - Hôpital COCHIN, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: This web link leads to the website of SAFIR, which is a French learned society dedicated to refractive and cataract surgery with implants. It contains an educational section on multifocal implants and cataract surgery to better understand the protocol. — https://www.safir.org/contenu-educatif-e-membre/